CLINICAL TRIAL: NCT00995813
Title: Pilot Study of the Safety and Immunogenicity of the Rotavirus Vaccine in Infants With Intestinal Failure
Brief Title: Pilot Study of the Rotavirus Vaccine in Infants With Intestinal Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Thrasher Research Fund (Other); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Patrick Javid, Principal Investigator, Seattle Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RS_Rota_vaccine_if
Record Dates: First submitted 2009-10-13; First posted 2009-10-15 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Intestinal Failure; Rotavirus Vaccines
Keywords: Intestinal failure; Rotavirus vaccine; Infants
MeSH Terms: conditions — Intestinal Failure | interventions — RIX4414 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Rotarix — A rotavirus vaccine (Rotarix) will be administered in two doses, 8 weeks apart, in infants between 6 and 14 weeks of age. The standard dosage is 1 mL administered orally or per gastrostomy tube.

SUMMARY:
The purpose of this study is to assess the safety and immune response of the rotavirus vaccine in infants who have undergone abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Infants with one of the following diagnoses:

  * necrotizing enterocolitis requiring operation;
  * congenital atresia of the intestine;
  * gastroschisis;
  * midgut volvulus requiring bowel resection; or
  * long-segment intestinal aganglionosis
* Minimum gestational age of 35 weeks at time of first vaccine dose

Exclusion Criteria:

* immunocompromise secondary to HIV infection or immunodeficiency state
* active use of corticosteroid or other immunosuppressive agents
* active infection as defined by fever > 38°C within 24 hours, positive blood culture within 7 days, or positive urine culture within 3 days of enrollment
* severe malnutrition as defined by serum albumin < 2.0 mg/dL or serum prealbumin < 6 mg/dL.

Ages: 6 Weeks to 14 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2009-12; Primary Completion 2012-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The safety of the rotavirus vaccine in infants with intestinal failure is the primary outcome variable. | 1-12 weeks following vaccine administration

SECONDARY OUTCOMES:
The secondary outcome measure is the preliminary measurement of the immunogenicity of the rotavirus vaccine in infants with intestinal failure. | 1-12 weeks following vaccine administration

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J Javid, MD, Principal Investigator — Seattle Children's Hospital and The University of Washington; Simon Horslen, M.B., ChB, Principal Investigator — Seattle Children's Hospital and The University of Washington; Janet Englund, MD, Principal Investigator — Seattle Children's Hospital and The University of Washington
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States